CLINICAL TRIAL: NCT00706069
Title: A Phase I Study Of Vinorelbine Oral Plus Capecitabine Combination In Patients With Metastatic Breast Cancer
Brief Title: Vinorelbine Oral Plus Capecitabine Combination In Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Nikos Malamos, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.06
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Vinorelbine oral; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vinorelbine oral plus Capecitabine
  Interventions: Drug: Vinorelbine oral; Drug: Capecitabine

INTERVENTIONS:
Drug: Vinorelbine oral — Vinorelbine at dose levels of 30mg, 40mg, 50mg, 60mg oral every Monday, Wednesday and Friday
  Other Names: Navelbine oral
Drug: Capecitabine — Capecitabine at dose levels of 800 mg/m2, 950mg/m2, 1100mg/m2, 1250mg/m2 per os from day 1 to day 14 every 21 days
  Other Names: Xeloda

SUMMARY:
This study will evaluate the toxicity and secondary the efficacy of the combination vinorelbine plus capecitabine in metastatic breast cancer patients

DETAILED DESCRIPTION:
The combination capecitabine-vinorelbine, with iv administration of vinorelbine, has been studied in a phase [I]/[II], with favourable profile of toxicity in pretreated patients with anthracyclines and/or taxanes (Oncology News International vol 12, no 3, suppl 2, 2003).

In a study of toxicity and effectiveness, Vanhopher reported objective response rates (PR) in 21 from 45 patients (47%) and stabilization of disease (SD) in 16 patients (36%). Severe leucopenia (grade 4), was reported in 5% of patients (Borquez D, et al: Proc Am Soc Clin Oncol 19: Abstract 420, 2000)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer
* Age 18-75 years
* Bidimensionally measurable or evaluable disease
* Performance status (PS) 0-2 (ECOG)
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide, or surgical sterilization) during treatment and for three months after completing treatment
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the UNL in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases); adequate renal function (serum creatinine <1.5 times the upper normal limit); and adequate bone marrow function(neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L)
* At least three weeks from completion of irradiation
* Life expectancy ≥ 12 weeks
* Patients able to take oral medication
* written informed consent

Exclusion Criteria:

* Active infection
* Brain metastases
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Malnutrition (loss of ≥ 20% of the original body weight)
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of vinorelbine oral plus capecitabine combination | Toxicity assessment at 1st cycle
Dose Limited Toxicity (DLT) of vinorelbine oral plus capecitabine combination. | Toxicity assessment at 1st cycle

SECONDARY OUTCOMES:
Response Rate | Response evaluation at 3rd and 6th cycle by CT's or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Malamos, MD, Principal Investigator — "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology
Locations (4):
- Greece (4):
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion